CLINICAL TRIAL: NCT06322134
Title: Incidence and Characteristics of Drowning Patients at Sea Treated by the Royal Danish Air Force's Search And Rescue Helicopters From 2014-2023: a Nationwide Registry-based Study
Brief Title: Drowning Incidents Treated by the Danish SAR Helicopters
Acronym: DROWN_SAR
Status: Completed | Type: Observational
Sponsor: Prehospital Center, Region Zealand (Other)
Collaborators: Danish Defence (Unknown)
Responsible Party: Principal Investigator, Niklas Breindahl, Principal Investigator, Region Zealand
Other Study IDs: DROWN_SAR
Record Dates: First submitted 2024-03-07; First posted 2024-03-20 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Drowning; Drown; Drowning; Anoxia; Drowning, Near; Drowning and Nonfatal Submersion; Drowning or Immersion of Unknown Intent; Drowning and Submersion, Undetermined Intent; Drowning and Submersion While in Natural Water; Drowning and Submersion Due to Sailboat Sinking; Drowning and Submersion Due to Fall Off Ship
Keywords: Drowning; Danish Drowning Formula; Royal Danish Air Force; Search And Rescue (SAR); Emergency Medical Service (EMS); Registry; Retrospective; Epidemiology; Danish Prehospital Drowning Data
MeSH Terms: conditions — Drowning; Hypoxia; Near Drowning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fatal drowning: Prehospital mortality following a drowning incident, defined as a dichotomous variable (dead or alive) evaluated at case termination. Patients admitted to the hospital with cardiac arrest were considered fatal drowning incidents in this study.
  Interventions: Other: Drowning incident
- Non-fatal drowning: Drowning incidents where the patient had spontaneous circulation at hospital admission.
  Interventions: Other: Drowning incident

INTERVENTIONS:
Other: Drowning incident — Patients categorized as drowning have been experiencing respiratory impairment from submersion or immersion in liquid and needing rescue by the Royal Danish Air Force's Search and Rescue (SAR) helicopters.

SUMMARY:
Improving oxygenation and ventilation in drowning patients early in the field is critical and may be lifesaving. This may be achieved by helicopter emergency medical services (HEMS) such as the Danish Air Ambulance, or the Royal Danish Air Force's Search And Rescue (SAR) helicopters. The SAR operates in all weather conditions and is equipped with a hoist system, able to hoist patients from the sea or small ships without helipads. This study aimed to estimate the incidence of drowning missions attended by the Royal Danish Air Force's SAR helicopter and describe patient characteristics and prehospital interventions.

DETAILED DESCRIPTION:
The national Danish Drowning Cohort contains data on all fatal and non-fatal drowning patients treated by the Emergency Medical Services. However, data on drowning patients treated by the SAR helicopters is reported in a separate system.

The population of drowning patients treated by the SAR helicopters has never been described, thus contributing to the potential underreporting of the most critically ill drowning patients in Denmark. Given the rarity of drowning, registry-based studies are needed to provide patient characteristics and evaluate critical care interventions performed on this group of patients.

This study aims to identify and describe a national cohort of drowning patients at sea treated by the Royal Danish Air Force's SAR helicopters from 2014 to 2023.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated by the Danish SAR helicopters AND
* Drowning as defined by the WHO (the process of experiencing respiratory impairment from submersion or immersion in liquid)

Exclusion Criteria:

* Patients who have not been immersed or submersed.
* Duplets.
* Interhospital transfers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Drowning patients will be identified through manual validation of the Royal Danish Air Force's SAR helicopter's records using the internationally accepted definitions of fatal and non-fatal drowning incidents.
  Drowning was defined by the WHO in 2002 as "the process of experiencing respiratory impairment from submersion or immersion in liquid".
  If the incident involved submersion or immersion, but the patient did not experience respiratory impairment, the incident was categorised as a water rescue.
Sampling Method: Non-Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Annual incidence of drowning treated by the Danish SAR helicopters from 2014-2023 | 1 year
  The incidence will be reported as the annual number of cases.
Annual incidence rate of drowning treated by the Danish SAR helicopters from 2014-2023 | 1 year
  The incidence rate as the annual number of cases per 100,000 person-years.

SECONDARY OUTCOMES:
Spatial distribution of drowning patients treated by the Danish SAR helicopters from 2014-2023 | The map will display all drowning incidents treated by the Danish SAR helicopters from 2014-2023.
  The spatial distribution of drowning incidents will be displayed on a map of Denmark, with each case presented with a single entry based on the geographical coordinates of the incident.

CONTACTS AND LOCATIONS:
Overall Officials: Helle Collatz Christensen, Ass. Prof., Study Director — Prehospital Center, Region Zealand
Locations (1):
- Prehospital Center, Næstved, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analysed during the current study are available from the corresponding author upon reasonable request.

REFERENCES:
- [Background] Breindahl N, Wolthers SA, Jensen TW, Holgersen MG, Blomberg SNF, Steinmetz J, Christensen HC; Danish Cardiac Arrest Group. Danish Drowning Formula for identification of out-of-hospital cardiac arrest from drowning. Am J Emerg Med. 2023 Nov;73:55-62. doi: 10.1016/j.ajem.2023.08.024. Epub 2023 Aug 15. PMID 37619443
- [Background] Breindahl N, Wolthers SA, Moller TP, Blomberg SNF, Steinmetz J, Christensen HC; Danish Drowning Validation Group. Characteristics and critical care interventions in drowning patients treated by the Danish Air Ambulance from 2016 to 2021: a nationwide registry-based study with 30-day follow-up. Scand J Trauma Resusc Emerg Med. 2024 Mar 6;32(1):17. doi: 10.1186/s13049-024-01189-y. PMID 38448994